CLINICAL TRIAL: NCT07213219
Title: Exploration of the Reward System in Parkinson's Patients With Paradoxical Sleep Behavior Disorders: a Multimodal Imaging Study
Brief Title: PET-MRI of Reward System in Parkinson's Disease With RBD
Acronym: RBD Impulse
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PHRC I 2022 BEAL; 2024-A00544-43 (Other: IDRCB)
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Parkinson's Disease (PD)
Keywords: Impulse Control Disorders; Rapid Eye Movement Sleep Behavior Disorder; Parkinson's Disease; Positron Emission Tomography; [¹¹C]raclopride; Magnetic Resonance Imaging
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; REM Sleep Behavior Disorder

STUDY DESIGN:
Intervention Model Description: Exploratory cross-sectional comparative study of pathophysiology. 2 groups will be compared :
  * MPI with RBD
  * MPI without RBD (control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPI with RBD (Experimental)
  Interventions: Other: PET-MRI (Positron Emission Tomography - Magnetic Resonance Imaging).
- MPI without RBD (Experimental): control group
  Interventions: Other: PET-MRI (Positron Emission Tomography - Magnetic Resonance Imaging).

INTERVENTIONS:
Other: PET-MRI (Positron Emission Tomography - Magnetic Resonance Imaging). — The PET-MRI will be performed using a Siemens Biograph mMR hybrid PET-MRI scanner. A 60-minute dynamic PET acquisition will begin following the intravenous injection of \[¹¹C]raclopride (a radiotracer agonist of dopamine D2/D3 receptors) synthesized in the radiopharmaceutical laboratories of CERMEP. Simultaneously with the PET acquisition, brain MRI sequences will be acquired: 3D anatomical T1 and 3D T2, SWI, diffusion MRI (DTI), resting-state functional MRI, and arterial spin labeling (ASL) perfusion MRI.
  Patients will undergo two PET-MRI scans on two consecutive days under two pharmacological conditions: Off and On dopamine:
  * Day 1:** The first PET-MRI session (TEPDopaOff) will be performed after a 12-hour withdrawal from usual dopaminergic treatment (Off dopamine).
  * Day 2:** The second PET-MRI session (TEPDopaOn) will be similar to the first, except it will take place 1 hour after administration of immediate-release Levodopa

SUMMARY:
Impulse control disorders (ICDs) are frequently observed in Parkinson's disease (PD) and can have a major functional impact on the quality of life of both the patient and their entourage. The primary risk factor for the emergence of ICDs in PD is long-term dopaminergic treatment, but other risk factors, such as rapid eye movement sleep behavior disorder (RBD), have recently been identified. The mechanisms leading to ICDs in PD remain debated, but it has been shown that the dopaminergic mesocorticolimbic pathways play a key role in reward, learning, and reinforcement processes, as well as in the regulation of impulsivity. PET studies using [11C]raclopride, a tracer that allows evaluation of the postsynaptic availability of dopamine D2/D3 receptors, have demonstrated abnormal sensitization of the mesocorticolimbic dopaminergic system (the reward system), particularly in the ventral striatum, in Parkinson's patients with ICDs when presented with appetitive stimuli or during gambling tasks. However, this has never been studied in patients with and without RBD. Parkinson's patients with RBD may present greater impairment of mesocorticolimbic pathways than those without RBD, particularly abnormal sensitization and postsynaptic modifications of the dopaminergic system, which could predispose patients to the emergence of ICDs when exposed to dopaminergic agonists. Confirming a particular pattern of denervation in Parkinson's patients with RBD that may favor the emergence of ICDs constitutes a personalized medicine approach with a readily identifiable risk marker in routine clinical practice and offers the possibility of adapting the management of these patients.

The main objective of this study is to investigate the availability of D2 dopaminergic receptors in subcortical structures (particularly the mesocorticolimbic system) in patients with idiopathic Parkinson's disease, depending on the presence or absence of RBD

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45 to 80 years
* Patients diagnosed with idiopathic Parkinson's disease (PD) according to the Movement Disorder Society criteria
* Disease duration between 3 and 7 years
* Patients receiving chronic dopaminergic treatment including levodopa for at least one year to avoid tolerance issues during acute levodopa administration
* Ability to cooperate and understand, allowing strict compliance with the conditions set forth in the protocol
* Patients affiliated with or beneficiaries of a social security system
* Volunteer patients capable of providing informed consent to participate in the research

Exclusion Criteria:

* Patients suffering from neurological disorders other than idiopathic Parkinson's disease (PD)
* Patients with severe depression (Beck Depression Inventory \[20] (BDI) score > 30), apathy (Starkstein scale \[21] score ≥ 14), cognitive impairment (Montreal Cognitive Assessment \[MoCA] \[22] score < 25), or impulse control disorders (QUIP - Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease \[23], score ≥ 1)
* Patients with severe motor symptoms: patients with an MDS-UPDRS III score > 45 will be excluded to avoid severe discomfort or interfering tremor (tremor item ≥ 3 in any body part) in the OFF state during PET-MRI acquisition. Patients with severe dyskinesias will also be excluded due to technical issues related to movement
* Patients under guardianship, curatorship, deprived of liberty, or under legal protection
* Pregnant or breastfeeding women
* Patients with contraindications to PET-MRI (e.g., those with pacemakers or insulin pumps, metallic prostheses or intracerebral clips, claustrophobia, neurosensorial stimulators or implantable defibrillators, cochlear implants, ferromagnetic ocular or cerebral foreign bodies near nervous structures, uncooperative or agitated patients, neurosurgical ventriculoperitoneal shunts, dental appliances)
* Refusal to participate

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
[¹¹C]raclopride binding potential (BP, unitless) measured with PET-MRI in mesocorticolimbic brain structures between participants with and without RBD, off treatment. | During MRI exploration (3 months after inclusion visit)
  The primary outcome measure corresponds to the Difference in binding potential (BP) of [¹¹C]raclopride in the brain structures of the mesocorticolimbic network between groups with and without RBD at baseline evaluation, off treatment, derived from PET-MRI imaging in mesocorticolimbic brain structures.
  The measurement tool is the [¹¹C]raclopride PET-MRI. BP is a unitless quantitative parameter (ratio between specifically bound radioligand and non-displaceable radioligand in tissue).

SECONDARY OUTCOMES:
[¹¹C]raclopride binding potential (BP, unitless) measured with PET-MRI in mesocorticolimbic brain structures between participants with and without RBD following acute administration of Levodopa | During MRI exploration (3 months after inclusion visit)
MDS-UPDRS III motor score | at the inclusion visit
  UPPS impulsivity scale score
Starkstein apathy scale score | at inclusion visit
BDI depression score | at inclusion visit
Ardouin Scale of Behavior in Parkinson's Disease) scores (hypodopaminergic and hyperdopaminergic items) | at inclusion visit
Total levodopa equivalent dose and for agonists (in mg/day) | at inclusion visit
Voxel-wise parametric statistical maps (SPM) across the whole brain comparing PET parametric images ([¹¹C]raclopride BP) | During MRI exploration (3 months after inclusion visit)
Voxel-wise parametric statistical maps (SPM) across the whole brain comparing MRI images. | During MRI exploration (3 months after inclusion visit)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte BEAL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU Clermont-Ferrand, Clermont-Ferrand,, Clermont-Ferrand
  - CH Le Puy en Velay, Le Puy-en-Velay